CLINICAL TRIAL: NCT00055159
Title: Treatment of Jugular, Subclavian, and/or Innominate Vein Thrombosis With Low Dose Recombinant Tissue Plasminogen Activator Plus Anticoagulation
Brief Title: Low-Dose rtPA to Treat Blood Clots in Major Arm or Neck Veins
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030113; 03-CC-0113
Record Dates: First submitted 2003-02-20; First posted 2003-02-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-12-10

CONDITIONS: Thrombosis
Keywords: RT PA; Blood Clots; Catheter Directed Thrombolytic Therapy; Alteplase; Deep Vein Thrombosis; DVT
MeSH Terms: conditions — Thrombosis; Venous Thrombosis

INTERVENTIONS:
Procedure: Pulse-sprayed injection of recombinant tissue plasminogen activator (rtPA)

SUMMARY:
This study will test the effectiveness of low-dose recombinant tissue plasminogen activator (rtPA, or alteplase) in dissolving blood clots in major arm or neck veins. rtPA is given to patients with heart attacks to dissolve blood clots in blocked coronary arteries. Blood clots that develop in major arm or neck veins usually develop after a venous access device (VAD) or catheter has been placed in the vein. The clot often causes arm, shoulder or neck swelling and pressure or discomfort. Current treatments include removing the VAD, using blood thinners such as heparin and warfarin, or using rtPA to dissolve the clot. All these options have disadvantages, however, including the risk of abnormal bleeding. This study will evaluate whether lower doses of rtPA can effectively dissolve clots without requiring an extended hospital stay, as is needed with the current higher-dose regimen.

Patients 18 years of age and older who are enrolled in or are being evaluated for a Clinical Center study and who have a blocked jugular, axillary, subclavian, or brachiocephalic vein may be eligible for this study. The blockage may or may not be associated with use of a VAD.

Participants will have one or two treatments with a low dose of rtPA, followed by a blood thinner taken by mouth or by injection for 5 to 7 weeks. On the first treatment day, the patient has a venogram, in which a catheter is placed in an arm vein and passed up to and through the blood clot that is blocking the blood flow in the vein. This is done under an x-ray machine so the radiologist can see exactly where the tube is going. Then, rtPA is injected into the clot about every 30 seconds for 15 to 30 minutes. The catheter is kept in place to maintain access to the vein for additional treatment the next day, if needed. The patient then begins treatment with heparin, either as an outpatient or an inpatient. A second venogram is done the next day. If the venogram shows that the vein is open, anti-clotting treatment with heparin or warfarin continues. If the venogram shows that the vein is still blocked, the rtPA treatment is repeated while the blood thinner treatment continues. The patient has a third venogram the following day. If the vein has opened, heparin and warfarin treatment continues. If the vein is still blocked, the patient's participation in the study ends. Although the patient is no longer formally in the study, he or she may choose to receive additional treatments with rtPA in higher doses at NIH or to continue using blood thinners under the direction of the primary physician.

Blood tests are done during blood thinning therapy to monitor and adjust the dosage. Additional blood samples are taken before and at timed intervals after each rtPA treatment to measure the response to therapy. Patients who benefit from rtPA treatment remain on blood thinners for 5 to 7 weeks and then return to NIH for a follow-up venogram to see if the vein is still open. During warfarin therapy, blood tests are done every few days during the first week or two and every 2 weeks thereafter to ensure the optimal drug dose is being administered. If the repeat venogram at 5 to 7 weeks shows that the vein has closed, the blood thinners (warfarin or heparin) will be stopped and the patient's participation in this study will end. If the vein has remained open, the patient's doctor will decide whether or not to continue anti-clotting therapy.

DETAILED DESCRIPTION:
Deep vein thrombosis of the central veins of the upper extremity and neck is most commonly seen at the Clinical Center as a consequence of use of central venous access devices (VADs) required for intravenous medication treatment programs at the NIH. In order to relieve discomfort associated with this condition or restore patency of the central veins, we successfully developed a treatment program employing intraclot pulse-sprayed injection of recombinant tissue plasminogen activator (rtPA) and anticoagulation with heparin plus warfarin (Protocol 95-CC-0053). Recent laboratory kinetic studies of thrombolysis with rtPA suggest that more rapid thrombolysis can be achieved with rtPA doses that are more than 10 times lower than the doses used in our earlier protocol. The purpose of this protocol is to evaluate whether these lower doses translate into more effective thrombolysis in the clinical setting, so that we may modify our thrombolysis treatment to make it more effective, potentially safer, and less costly than our previous protocol. This proposed protocol still utilizes pulse spray injection of rtPA directly into the thrombus as before, but evaluates the efficacy and safety of using a total of 4 mg or less of rtPA each day for thrombolytic therapy. As this lower dose of rtPA has been found to be safe in catheter clearance applications, hospitalization will not be required as part of the protocol. Patients who elect to have this procedure performed as outpatients will also receive anticoagulation with standard regimens using subcutaneous low molecular weight heparin (LMWH) alone, or with gradual conversion to oral warfarin.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adults (18 years or older) are eligible for this study.

Patients must be enrolled in or actively being evaluated for a protocol at the Clinical Center.

Patient must be able to give informed consent and be able to follow anticoagulation regimen if enrolled.

Occlusive thrombosis of jugular, axillary, subclavian, or brachiocephalic veins must be documented by ultrasound, or venography (Occlusive meaning complete blockage of blood flow across affected venous segment). Although most thrombi will be associated with a VAD, this is not a requirement.

Estimated duration of thrombosis should not exceed 4 weeks based on clinical history.

Postpartum mothers are eligible for this treatment, but nursing mothers will be instructed to refrain from breast feeding their infants for 24 hours after each venogram or contrast study.

EXCLUSION CRITERIA:

Pregnancy: Although the abdomen can be shielded from medical radiation required for the procedures, the use of contrast media, thrombolytic enzymes, and anticoagulation can potentially have adverse effects on a pregnancy, so that thrombolytic therapy is contraindicated during pregnancy.

Children are excluded from this protocol but are eligible for the high dose regimen that is the current standard at NIH.

Patients who are cognitively impaired and cannot give consent will not be eligible for this protocol. The current high dose regimen remains an option, if appropriate consent can be obtained from legally responsible guardian or family member.

Patients with known diabetic or other retinopathy will be excluded unless cleared for treatment by an ophthalmologist.

Gastrointestinal or internal bleeding (except microscopic hematuria) within the previous two weeks; active peptic ulcer disease; familial or acquired bleeding diathesis not attributable to heparin administration (prothrombin time greater than 14 s, APTT greater than 35s, fibrinogen less than 150mg/dl); thrombocytopenia less than 50,000 microliters.

History of cerebrovascular accident or neurosurgery within previous 2 months

Lumbar puncture within previous 2 weeks, or patients with epidural catheters, current or in the past 2 weeks.

Major surgery, trauma, or deep organ biopsy within the previous 10 days: recent onset (less than 10 days) of atrial fibrillation without anticoagulation, Known right to left cardiac shunts, and pulmonary arteriovenous malformations.

Severe hypertension (systolic pressure greater than 200 mmHg, diastolic pressure 110 mmHg)

Renal insufficiency with serum creatinine greater than 2.5mg/dl

History of anaphylactic reaction to iodinated contrast material.

History of heparin-induced thrombocytopenia.

Acute Pericarditis

Known defect of cardiac septum with right to left intracardiac shunt.

Pulmonary arteriovenous malformation.

Bacterial endocarditis.

Intracranial neoplasm, arteriovenous malformation, and aneurysm with evidence, clinically or by imaging, of hemorrhage in previous 2 months excludes participation. If there has been no evidence of bleeding, these patients can be considered for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-02-19; Study Completion 2007-12-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Turpie AG, Levine MN, Hirsh J, Ginsberg JS, Cruickshank M, Jay R, Gent M. Tissue plasminogen activator (rt-PA) vs heparin in deep vein thrombosis. Results of a randomized trial. Chest. 1990 Apr;97(4 Suppl):172S-175S. PMID 2108855